CLINICAL TRIAL: NCT02742207
Title: Evaluation of Renal Function and Fluid Balance of Patient Undergoing Electrical Cardioversion for Atrial Fibrillation
Brief Title: Renal Function Post Cardioversion for Atrial Fibrillation
Acronym: AFCARD-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Dan Gilon, Director, Non-Invasive Cardiology/Echocardiography, Hadassah Medical Organization
Other Study IDs: HMO-15-0645
Record Dates: First submitted 2016-04-09; First posted 2016-04-18 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Renal Insufficiency; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: All comers with Atrial fibrillation
  Interventions: Other: Electrical atrial fibrillation Cardioversion; Other: Cardioversion

INTERVENTIONS:
Other: Electrical atrial fibrillation Cardioversion — Electrical cardioversion for patients admitted for Atrial Fibrillation
  Other Names: Cardioversion
Other: Cardioversion — Electrical cardioversion for patients admitted for Atrial Fibrillation

SUMMARY:
Atrial fibrillation is a common arrhythmia which requires electrical cardioversion in many patients in order to regain sinus rhythm. In a previous retrospective study a complication of acute renal failure was found in 17% of the patients after cardioversion.(The incidence and prognosis of renal dysfunction following cardioversion of atrial fibrillation. Helman Y,...Gilon D et al:Cardiology 2013;124(3);184-9.) Another complication previously described after cardioversion is pulmonary edema.

In this prospective study the investigators aim to evaluate the risk of acute renal failure post cardioversion. In addition the investigators would like to evaluate hemodynamic changes, fluid balance and sodium levels in patients post cardioversion as a potential mechanism for both acute renal failure and pulmonary edema post cardioversion. In order to assess hemodynamic changes the investigators will use a non-invasive FDA approved device called NICaS (Non-Invasive Cardiac System). This system calculates cardiac output, cardiac index and peripheral vascular resistance in a non-invasive, fast and accurate way.

ELIGIBILITY:
Inclusion Criteria:

* All patients with new onset atrial fibrillation

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with new onset atrial fibrillation. Meaning less than three days.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Renal dysfunction | Short term - One month
  Creatinine Clearance less 25 percent.

SECONDARY OUTCOMES:
Mortality | One year
  Death

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hellman Y, Cohen MJ, Leibowitz D, Loncar S, Gozal D, Haviv YS, Haber G, Afifi M, Rosenheck S, Lotan C, Pollak A, Gilon D. The incidence and prognosis of renal dysfunction following cardioversion of atrial fibrillation. Cardiology. 2013;124(3):184-9. doi: 10.1159/000346618. Epub 2013 Mar 9. PMID 23485988